CLINICAL TRIAL: NCT05648955
Title: Muscle Mass in Patients With Colorectal or Lung Cancer When Receiving an Oral Nutritional Supplement During Anti-cancer Treatment
Brief Title: Effect of an Oral Nutritional Supplement on Muscle Mass During Anticancer Treatment
Acronym: ALLIES
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MPR15ON89540
Record Dates: First submitted 2022-08-10; First posted 2022-12-13 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer (CRC); Non-small Cell Lung Cancer (NSCLC)
Keywords: Muscle mass; oral nutritional supplement; colorectal cancer; non-small cell lung cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): An enriched high protein and high energy oral nutrition supplement (ONS)
  Interventions: Dietary Supplement: an enriched high protein and high energy oral nutrition supplement (ONS)
- Control product (Active Comparator): standard isocaloric high energy normal protein isocaloric ONS
  Interventions: Dietary Supplement: an enriched high protein and high energy oral nutrition supplement (ONS)

INTERVENTIONS:
Dietary Supplement: an enriched high protein and high energy oral nutrition supplement (ONS) — NA (see intervention name)

SUMMARY:
Malnutrition and low muscle mass (sarcopenia) are common problems in patients with cancer. However, a low muscle mass is associated with negative clinical outcomes in patients with cancer. Therefore, it is very important to maintain muscle mass in this population. This study aims to investigate the effect of an oral nutritional supplement on skeletal muscle mass during anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III or IV colorectal or non-small cell lung cancer
* Scheduled for the first cycle of any line of a systemic treatment: chemotherapy, concurrent chemoradiotherapy, immunotherapy or targeted treatment with a planned duration of at least 9 weeks
* Performance status Eastern Cooperative Oncology Group (ECOG) score 0 or 1
* Age ≥ 18 years

Exclusion Criteria:

* Weight loss >10% in the last 6 months
* Body Mass Index > 30.0 kg/m2
* Life expectancy < 3 months
* Receiving enteral (tube) or parenteral nutrition
* Presence of ileostoma or ileal pouch (except for an ileostomy at or near the terminal ileum which does not affect absorption of nutrients other than sodium, potassium, and water, in the opinion of the investigator)
* Allergy to cow's milk protein, soy or fish, requiring a fibre-free diet or suffering galactosemia or lactose intolerance
* Known pregnancy or lactation
* Current alcohol or drug abuse in the opinion of the investigator
* Wearing an electronic implant and/or pacemaker
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within 14 days prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cross-sectional skeletal muscle mass area on the third vertebral level (L3) [cm2] | 12 weeks
  between baseline and after 12 weeks of intervention as measured with a CT scan, between the two interventions

SECONDARY OUTCOMES:
Change in health-related quality of life as measured with the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30 global health score) | ~13 weeks
  between baseline and end of study [score], between the two interventions.

OTHER OUTCOMES:
Change in health-related quality of life as measured with the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30 global health score) | ~13 weeks
  between baseline and end of study
Inflammation status | ~13 weeks
  at baseline, visit 2, visit 3 and end of study (visit 5):
  * Neutrophil/lymphocyte ratio
  * CRP [mg/L]
  * Albumin [g/L]
  * Modified Glasgow Prognostic Score (mGPS) [score 0/1/2]
    * CRP ≤ 10 mg/L and albumin ≥ 35 g/L or CRP ≤ 10 mg/L and albumin < 35 g/L -> score 0
    * CRP > 10 mg/L and albumin ≥ 35 g/L -> score 1
    * CRP > 10 mg/L and albumin < 35 g/L -> score 2
Change in performance status ECOG | ~13 weeks
  between baseline and end of study [score]
Change in physical function | ~13 weeks
  between baseline and end of study: 30 seconds chair stand test [number]

CONTACTS AND LOCATIONS:
Locations (1):
- UCC, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No